CLINICAL TRIAL: NCT07327294
Title: An Open-label, Multicenter Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of XNW34017 in Patients With Advanced Solid Tumors
Brief Title: A Phase I/II Study to Evaluate XNW34017 in Patients With Advanced or Metastatic Solid Tumor
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Evopoint Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XNW34017-I/II-01
Record Dates: First submitted 2025-12-12; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XNW34017 (Experimental)
  Interventions: Drug: XNW34017

INTERVENTIONS:
Drug: XNW34017 — Drug Name: XNW34017 Tablets Dosage Form: Tablet Strength: 5 mg, 50 mg Route of Administration: Oral Storage Instructions: Store in a sealed container, protected from light, at temperatures not exceeding 30°C.

SUMMARY:
This study is an open-label, dose-escalation, multicenter Phase I/II study conducted in patients with advanced solid tumors. The target population for this study consists of patients with advanced solid tumors who have failed or are intolerant to standard treatments. The study is divided into two parts: the dose-escalation phase and the dose-expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Dose escalation phase: Subjects with advanced and/or metastatic malignant solid tumors who have failed standard treatment or lack effective standard treatment, and have histologically or cytologically confirmed diagnosis.
2. Dose expansion phase, including but not limited to: Advanced and/or metastatic small cell lung cancer, prostate cancer, etc., with disease progression confirmed by histopathology, and failure in the following anti-cancer treatments:

   Small cell lung cancer: Patients with small cell lung cancer who have progressed or relapsed after receiving at least two prior systemic treatment regimens.

   Metastatic castration-resistant prostate cancer (mCRPC): Patients who have previously received treatment with enzalutamide or abiraterone and have experienced disease progression. At screening, serum testosterone should be at castration levels (≤ 50 ng/dL or ≤ 1.73 nmol/L). For patients who have not undergone bilateral orchiectomy, LHRHa therapy should be administered ≥ 4 weeks prior to the first dose of study treatment and continued throughout the study.
3. The subject must be ≥ 18 years of age at the time of signing the informed consent.
4. At least one measurable lesion according to RECIST 1.1 criteria (applicable to the backfill cohort and dose expansion phase).
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1.
6. The subject's organ function levels must meet the following requirements within 7 days prior to the first dose:

   Absolute Neutrophil Count (ANC) ≥ 1.5×10^9/L, Platelet Count ≥ 100×10^9/L, Hemoglobin ≥ 90 g/L; Creatinine Clearance ≥ 60 ml/min (calculated using the Cockcroft-Gault formula) or Serum Creatinine (Cr) ≤ 1.5 times the upper limit of normal; Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) levels ≤ 2.5 times the upper limit of normal (ULN), for liver cancer/liver metastasis patients, AST/ALT should be ≤ 5×ULN; Total Bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN), for patients with Gilbert's Syndrome, Direct Bilirubin (DBIL) must be ≤ 2×ULN; International Normalized Ratio (INR) ≤ 1.2 (without anticoagulant treatment), Activated Partial Thromboplastin Time (APTT) ≤ 1.25×ULN; for subjects who have been on stable-dose anticoagulant therapy (e.g., warfarin) for ≥8 weeks, INR must be ≤3.
7. Life expectancy ≥ 12 weeks.
8. Female participants of childbearing potential must undergo a urine or serum pregnancy test within 7 days prior to starting the study medication, and the result must be negative. If the urine pregnancy test is positive or inconclusive, a serum pregnancy test must be performed.
9. During the study and for 6 months after the last dose of the study drug, an effective, medically approved contraception method (e.g., intrauterine device, contraceptive pills, or condoms) must be used. For male participants with a female partner of childbearing potential, they must either be surgically sterilized or agree to use an effective contraception method during the study and for 6 months after the last dose of the study drug. Additionally, male participants must agree not to donate sperm throughout their study participation and for at least 6 months after their last dose of study drug.
10. The participant has given informed consent and has signed the informed consent form, and is willing and able to comply with the study procedures required by the protocol.

Exclusion Criteria:

1. Individuals who have had an allergic reaction to any component of the XNW34017.
2. The washout period of prior antitumor treatments before the first study drug treatment is insufficient, defined as follows:

   Chemotherapy, small molecule targeted therapy, or endocrine therapy < 2 weeks or 5 half-lives, whichever is shorter; Monoclonal antibody therapy < 3 weeks; Brain radiotherapy < 2 weeks, palliative radiotherapy < 2 weeks, curative radiotherapy < 4 weeks.
3. Subjects with double primary malignant tumors, except for the specific cancer being studied in this trial and any previously cured local tumors: non-invasive basal cell carcinoma or squamous cell carcinoma, non-invasive superficial bladder cancer, and any other tumors with a complete remission (CR) lasting more than 5 years.
4. Receiving a live vaccine within 4 weeks prior to the first study drug treatment. Note: Seasonal flu vaccines are generally inactivated vaccines and can be used; however, intranasal flu vaccines, which are live attenuated vaccines, are not permitted.
5. Use of granulocyte colony-stimulating factor (G-CSF) or granulocyte/macrophage colony-stimulating factor within 1 week prior to the first study drug treatment, or use of pegylated G-CSF within 2 weeks prior to the first study drug treatment. Receiving blood transfusion treatment within 2 weeks prior to the first study drug treatment. Use of erythropoietin (EPO) or IL-11 within 1 week prior to the first study drug treatment.
6. Subjects who have not yet recovered from the toxicity of prior anticancer treatments to CTCAE grade ≤ 1 or a stable condition, except for AEs that are not considered to pose a safety risk (e.g., hair loss).
7. A history of intracranial arteriovenous malformation, cerebral aneurysm, or stroke (including transient ischemic attack within 1 month prior to screening, but excluding old cerebral infarction and asymptomatic cerebral infarction).
8. Presence of any of the following hematologic risk factors:

   Known coagulation defects leading to an increased risk of bleeding; Diffuse alveolar hemorrhage caused by vasculitis; Persistent major bleeding; Trauma resulting in an increased risk of life-threatening bleeding; A history of severe extracranial injury or intracranial surgery within 8 weeks prior to the start of the trial.
9. Unable to provide tumor tissue samples for biomarker expression testing (for subjects unable to provide tissue samples, enrollment may be determined through consultation between the investigator and the sponsor).
10. Presence of clinically significant cardiovascular or cerebrovascular diseases:History of unstable angina;Myocardial infarction within 6 months prior to screening;Underwent angioplasty or coronary stent treatment within 6 months prior to screening;History of congestive heart failure with New York Heart Association (NYHA) classification of 3 - 4;Baseline QTc interval abnormality (QTcF > 450 ms);Occurrence of ≥ grade 2 ventricular arrhythmia within 6 months prior to screening;Poorly controlled hypertension: systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg despite standard antihypertensive treatment;Presence of cardiac disease/history that results in left ventricular ejection fraction (LVEF) < 50%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of AEs and SAEs | 24 months
  The incidence and severity of AEs and SAEs
ORR | 24 months
  ORR assessed by investigator

SECONDARY OUTCOMES:
Plasma concentrations of XNW34017 | 8 months
  Plasma concentrations of XNW34017
DCR | 24 months
  Disease control rate (DCR)
DOR | 24 months
  Duration of Response (DOR)
PFS | 24 months
  Progression Free Survival (PFS)
OS | 24 months
  Overall Survival(OS)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No